CLINICAL TRIAL: NCT06932731
Title: The Effects of Mind-Body Intervention Versus Befriending Intervention on Loneliness for Older Adults in Long-term Care: A Randomised Controlled Trial
Brief Title: Mind-Body Intervention for Older Adults in Long-term Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Szeto Cheuk Yan, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW 25-016
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Long Term Care Facility
Keywords: loneliness; mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mind-Body Intervention Group (Experimental): The entire intervention will be conducted in a group setting for 5 sessions. Each session 45 to 60 minutes weekly. Intervention is led by a registered nurse. Participants will be instructed to perform mind-body intervention during session and encouraged to have home practice between the next session.
  Interventions: Behavioral: Mind-body Intervention
- Befriending Intervention Group (Active Comparator): This group will receive befriending intervention provided by volunteers with health care background. Volunteers are either studying or graduated from a health science related programme. Participants will meet volunteers each week in a group setting for 5 sessions. Each session 45 to 60 minutes.
  Interventions: Behavioral: Befriending Intervention

INTERVENTIONS:
Behavioral: Mind-body Intervention — The Mind-Body Intervention group designed to included several elements with mind and body involvement such as mindful breathing, body scan, stretching, mindful movement as well as adapting mindful practice in their routine. Mind-Body Intervention group will join the activities in a group setting for 5 sessions. Each session 45 to 60 minutes. Intervention is led by a registered nurse. Each session (except for the first session) will start by sharing of practice from the past week. Followed by mind-body practices. Before the end of session, a group discussion on the practice of that day and reflection will be done.
  Arms: Mind-Body Intervention Group
Behavioral: Befriending Intervention — In this group, volunteer will spend time with the participants, engaging in conversation and join their routine activities by the time of visit or other scheduled activities in the institution (such as arts and crafts, playing board games or reminiscing activities).
  Arms: Befriending Intervention Group

SUMMARY:
Loneliness is a global health issue, particularly affecting the physical and mental health of older adults residing in long term care. The COVID-19 pandemic has further exacerbated isolation in these settings, calling for an urgent attention for finding an effective intervention to alleviate loneliness among long term care residents. Mind-body interventions (MBIs) present as a potentially promising approach aimed at reducing loneliness and mental wellbeing. This study aims to examine the effect of a nurse-led MBI compared to a befriending intervention on loneliness, quality of life, depression and level of mindfulness among older adults in long term care. The primary outcome is loneliness while secondary outcome is quality of life, depression and level of mindfulness.

DETAILED DESCRIPTION:
Loneliness is becoming a global health threat particularly in older population due to natural life events such as illness, death of a spouse and a lack of friends In Hong Kong, it has been reported the 58.1% of the older people experienced a high level of loneliness. Loneliness can have a devastating impact on mental and physical health by increasing the risk of dementia, depression, anxiety, stroke, myocardial infarction and poor quality of sleep.The associated mortality rate can be as high as 26% which is comparable to the harm of prime health dangers like alcohol and cigarette. The problem is particularly pressing for the older adults residing in long term care facilities during the COVID-19 pandemic. Outbreaks occurred in more than 90% of long-term care facility in Hong Kong. Resulting in further isolation in their own facilities or community isolation facilities. Preventing institutionalized older adults from being trapped in loneliness is of key importance. A promotion of intervention that is driven by theoretical framework and suitable for long-term care setting is required.

Mind-body practice has been extensively studied in different population such as chronic pain, heart disease, respiratory disease and community dwelling older adults. However, there is little evidence of wellbeing and loneliness reduction in mind-body practice among long term care older adults. This study will adopt befriending intervention as the control group. As befriending intervention is common in Hong Kong by volunteer visiting.

This study describes a randomised controlled trial designed to compare the effectiveness of a nurse-led MBI versus befriending intervention for LTC residents to reduce loneliness and enhance wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Long-term care residents aged 60 or above
* Communicable in Cantonese/Chinese
* Mentally competent (Abbreviated Mental Test score >6)
* Could read, write and understand Chinese language
* Able to provide written consent

Exclusion Criteria:

* Have regular practice of mindfulness once a week or more during the past 6 months
* Have any other contraindication or severe comorbidity that may limit their full participation (e.g. acute psychiatric conditions, severe hearing, vision impairment, or severe medical condition etc).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Loneliness | Baselines , 5 weeks, and 12 weeks after baseline
  For Mind-Body Intervention group and Befriending Intervention group, measured by UCLA 8-item Loneliness Scale is the shortened version of UCLA Loneliness Scale. The shortened scale consists of 8 questions with 4-point Likert scale ranged from 'never' to 'often'. The higher the score, the higher the level of perceived loneliness. Item 3 and Item 5 are reversely scored. Higher the score, the higher loneliness level.

SECONDARY OUTCOMES:
Level of mindfulness | Baselines , 5 weeks, and 12 weeks after baseline
  For Mind-Body Intervention group and Befriending Intervention group, measured by Multidimentional Assessment of Interoceptive Awareness (MAIA). It is a 32 items state-trait self reported questionnaires and is categorized into eight scales in 6 point Likert scale from 0 (never ) to 5 (always). A higher score indicates a more appraised interoceptive awareness and higher level of mindfulness.
Depression | Baseline, 5 weeks, and 12 weeks after baseline
  For Mind-Body Intervention group and Befriending Intervention group, measured by Geriatric Depression Scale 4 items (GDS-4) is a brief version of Geriatric Depression Scale 30 items (GDS-30). GDS-4 consists of 4 items from the original items of GDS-30. Total scores more than 2 is considered at risk of depression.
Health-related quality of life | Baseline , 5 weeks, and 12 weeks after baseline
  For Mind-Body Intervention group and Befriending Intervention group, measured by World Health Organization Well-Being Index (WHO-5 scale). It is a five items 6-point Likert-type scale from 0 (at no time) to 5 (all of the time). It focuses on positive emotions that included 5 items: "I have felt cheerful and in good spirits", "I have felt calm and relaxed", "I have felt cheerful and in good spirits", "I woke up feeling fresh and rested" and "I have felt active and vigorous". The participants are asked how well each of the items applied to them in the past two weeks. The higher the score, the better the mental wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Jojo Yan Yan Kwok, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, LKS Faculty of Medicine, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this study are available upon request from the principal investigator, Ms Szeto. These data are not publicly available, as they contain information that could compromise the privacy of research participants.